CLINICAL TRIAL: NCT00320970
Title: Angiotensin II Antagonism of TGF-Beta 1: A Candesartan Dose - TGF-Beta 1 Response Relationship Study
Brief Title: Angiotensin II Antagonism of TGF-Beta 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HI831
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2007-08-02 (Estimated); Status verified 2006-03

CONDITIONS: Diabetic Nephropathy; Hypertension
Keywords: TGF-Beta 1; Angiotensin II; Advanced glycation end products
MeSH Terms: conditions — Diabetic Nephropathies; Hypertension; Camurati-Engelmann Syndrome | interventions — candesartan

INTERVENTIONS:
Drug: Candesartan

SUMMARY:
Diabetic nephropathy is a frequent microvascular complication that occurs in approximately 40% of patients with either type 1 or type 2 diabetes. The most common cause of end-stage renal disease (ESRD) in the United States and in the developed world is diabetic nephropathy. Currently, more than half the United States ESRD population has diabetes. More effective therapies to prevent and treat diabetic nephropathy are urgently needed. One way to increase therapeutic effectiveness is to refine treatment targets based on improved understanding of how treatments modulate disease processes. The purpose of this study is to determine whether a treatment for diabetic nephropathy, the angiotensin receptor blocker candesartan, modifies mediators of kidney injury independent of blood pressure and the relationships to drug dose.

DETAILED DESCRIPTION:
Transforming growth factor-beta 1 (TGF-beta 1) is a potent inducer of extracellular matrix production and of fibrogenesis and has been associated with the occurrence of diabetic micro- and macrovascular complications. Several in vitro and in vivo studies have implicated TGF-beta 1 in the pathogenesis of diabetic kidney disease. Recent animal and in vitro experiments have demonstrated that ACE inhibitors and Angiotensin II (AT-II) receptor antagonists, including candesartan, decrease the synthesis and secretion of renal TGF-beta 1 and prevent the development of glomerulosclerosis, interstitial fibrosis, and progressive renal dysfunction. These protective effects appear to be unrelated to the antihypertensive effects of the agents.

Limited data in humans have supported these findings in patients with diabetic nephropathy. A recent human study with the AT-II receptor antagonist losartan demonstrated that the ability to correct microalbuminuria was independent of blood pressure control and correlated with normalization of circulating levels of TGF-beta 1. The results were further supported by the observation that markers of collagen type 1 metabolism were normalized in hypertensives in whom TGF-beta 1 was normalized with treatment but remained unaltered in the remaining hypertensives despite blood pressure control. Such findings are consistent with the recent observation that the AT-II receptor antagonist irbesartan is renoprotective independently of its blood pressure-lowering effect in patients with type 2 diabetes and microalbuminuria.

The use of ACE-inhibitors and AT-II receptor antagonists as a means to reduce progression of renal fibrosis is becoming increasingly widespread. Dosage recommendations to achieve this goal are unclear prompting some experts to ask whether TGF-beta 1 rather than blood pressure should be a therapeutic target. Although not verified under chronic conditions, previous short-term studies with the AT-II antagonist candesartan have demonstrated different dose-response relationships to exist for blood pressure, renal plasma flow, and plasma renin activity. It is likely that dose-response relationship differences also exist between the aforementioned parameters (particularly blood pressure) and TGF-beta 1. In type 1 diabetic patients treated with captopril a relationship was demonstrated between percent change in plasma TGF-beta 1 and percent decline in GFR. In another study of 21 patients with a baseline GFR of <75 ml/min there was a striking correlation between the captopril-induced reduction in serum TGF-beta 1 and 2-year change in GFR (r = -0.73, p =0.0001). This latter observation is particularly important in demonstrating that the relationship between TGF-beta 1 and rate of decline in kidney function can be modified through pharmacologic intervention.

The dosage range for candesartan according to the FDA approved package insert is 4 to 32 mg daily, adjusted based on blood pressure response. Whether the dose that effectively lowers blood pressure is sufficient to suppress urinary TGF-beta 1 concentrations is unknown. In the absence of data, many experts are already suggesting doses higher than needed to control hypertension. Including a maximum dose of candesartan 64 mg in a dose titration scheme will be important to help resolve this issue. Furthermore, it is unclear if the candesartan dose/concentration - effect relationship for TGF-beta 1 and blood pressure are dissimilar. Information regarding the relationship between candesartan dose and effect on urinary TGF-beta 1 concentrations in patients with diabetic nephropathy would be valuable in tailoring therapy and enhancing our understanding of the optimal use of agents that modulate the renin-angiotensin system.

Recent data in experimental models of diabetes indicate that the renin angiotensin system interacts with advanced glycation end products (AGEs) to produce kidney damage in diabetes. ACE inhibition in diabetic rats reduced circulating and renal accumulation of AGEs, possibly by increasing expression of the soluble receptor for AGEs. In a rat model of normoglycemia with AGE infusion, increased kidney expression of renin angiotensin system components along with structural changes similar to those in diabetic models was observed. Renin angiotensin system activation and kidney structural changes were reversed by valsartan. Therefore, modulation of AGEs may also be an important mechanism of kidney protection by renin angiotensin system inhibition in diabetes. This hypothesis is unexplored in humans. An exploratory sub-study will assess whether candesartan reduces urinary excretion of carboxymethyllysine, a prominent AGE, in patients with diabetic nephropathy.

Study Objectives and Hypotheses:

The overall objective of this study is to provide information that will improve kidney health in patients with diabetes. In a population of patients with type 2 diabetes, nephropathy, and hypertension the following hypotheses will be tested:

1. Changes in parameters of blood pressure, urinary TGF-beta 1, serum AT-II, and urinary albumin demonstrate correlation with changes in chronic candesartan dose and serum concentrations.
2. The candesartan dose and concentration response curves for BP and urinary TGF-beta 1 are significantly different and not predictive of one another.
3. Candesartan treatment will reduce urinary excretion of carboxymethyllysine.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Nephropathy (proteinuria >500 mg/day)
* Chronic Hypertension (as determined by current antihypertensive therapy and/or an average of diastolic blood pressure greater than 90 mmHg or greater or systolic blood pressure of 140 mmHg confirmed on at least two subsequent visits over one week or more).

Exclusion Criteria:

* Conditions associated with elevated TGF-Beta (e.g. rheumatoid arthritis, cancer, etc.).
* Conditions associated with alterations in serum levels of PIP and/or CITP (liver cirrhosis, osteoporosis, hyperthyroidism, multiple myeloma, osteolytic metastases, and systemic glucocorticoid treatment
* History of Stage III hypertension (diastolic BP > 110 mmHg or systolic BP > 180 mmHg) or a history of hypertensive urgency or emergency.
* NYHA Class III or IV heart failure
* Calculated creatinine clearance of less than 30 ml/min or serum creatinine > 3 mg/dL
* HbA1c > 10%
* Patients unable to be withdrawn for 2 weeks from AT-II antagonist or ACE- inhibitor therapy
* Blood Pressure <140/90 is unachievable in the absence of an AT-II antagonist or ACE-inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2002-08; Study Completion 2004-09

PRIMARY OUTCOMES:
Blood pressure
Urinary TGF-Beta 1
Serum angiotensin II
Urinary albumin
Urinary carboxymethyllysine

CONTACTS AND LOCATIONS:
Overall Officials: Katherine R. Tuttle, MD,FASN,FACP, Principal Investigator — Providence Medical Research Center
Locations (1):
- Providence Medical Research Center, Spokane, Washington, United States